CLINICAL TRIAL: NCT04270357
Title: Surgical Practices During Cholecystectomy in Algeria: Results of a Survey
Brief Title: Surgical Practices in Algeria : the Cholecystectomy
Status: Completed | Type: Observational
Sponsor: University of Oran 1 (Other)
Responsible Party: Principal Investigator, Anisse Tidjane, Maitre de conference grade A, University of Oran 1
Other Study IDs: UOran1
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: General Surgery; Cholecystectomy; Practice Guidelines as Topic
Keywords: cholecystectomy; middle income country; gallbladder; laparoscopy
MeSH Terms: interventions — Cholecystectomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cholecystectomy — Cholecystectomy is the surgical removal of the gallbladder. Cholecystectomy is a common treatment of symptomatic gallstones and other gallbladder conditions

SUMMARY:
An anonymous national survey involving all practicing Algerian surgeons was conducted. At the end of the survey, all data were captured and processed using the SPSS v20 software; χ 2 tests were used to compare different groups of surgeons.

DETAILED DESCRIPTION:
An anonymous national survey involving all practicing Algerian surgeons was conducted, this survey started the 1st November 2016 and ended the 1st September 2017.

Any digestive , general and visceral surgeon practicing in Algeria was eligible for this survey, surgeons in training "residents" and Algerian surgeons exercising overseas was systematically excluded.

The aim was to analyse some practice in accordance with the recommendations of the Society of American Gastrointestinal and Endoscopic Surgeons who published a guideline in 2010.

This elaborated form was an electronic one; it was performed using the open electronic platform "Google Form", the conception of the form was made by A.Tidjane "surgeon" and he was the first participant to this survey, considering his participation he was excluded from the seizure of the data. The analysis and interpretation of data was made by S.Benilha "bio-statistician", B.Tabeti "surgeon" and A.Tidjane.

The form consisted of two parts, the first concerning the surgeon's Wilaya of exercise, the rank of health structure of practice, his professional position , and the year of his graduation , the second part concerning his practices during the performing CH and the questions concerned the use of laparoscopy or open surgery to perform CH, the number of Trocars used, the technique to access the peritoneal cavity, the surgical technique, the use of intraoperative cholangiography "IOC", the technique of extraction of the gallbladder, systematic gallbladder macroscopic and histological examination, the systematic abdominal cavity drainage, systematic use of postoperative antibiotic prophylaxis, and the optimal duration of postoperative stay in the case of optimal patient with no preoperative incident or postoperative complication. At the end of the survey a question was asked to surgeons about the occurrence during their professional practice of an operative bile duct injury.

The language of instruction of surgeons in Algeria is French; the French was used to draft this form. This electronic form was distributed by email to all surgeons in the authors Mail lists, those first contacted surgeons had the mission not only to participate in this survey but also had the mission of distributing the electronic form to their surgeon colleagues. All incomplete responses were excluded.

Statistical analyses:

At the end of the survey, all data were captured and processed using the SPSS v20 software (IBM Inc., Chicago, IL, USA), a χ 2 tests were used to compare some surgical practices in different groups of surgeons, a (P < 0.05) was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* visceral an general surgeons practicing in Algeria.

Exclusion Criteria:

* surgeon under training.
* Algerian surgeon practicing abroad.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: any surgeon practicing in Algeria is subject to this survey. THE surgeons in Algeria are holders of a "DEMS or equivalent" diploma which authorizes them to perform surgery in Algeria.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Influence of surgeons caracteristics on surgical practices | 11 months
  The variables measured were of two types:
  A - linked to the characteristics of the surgeon participating in the survey:
  * Exercice place.
  * Type of exercise structure.
  * Grade of surgeon.
  * Date of graduation.
  * Weekly volume of surgery.
  * Use of laparoscopic surgery.
  B- Related to the surgeon's own practices when he performs this surgery:
  * Laparoscopic or open cholecystectomy.
  * Respect for the different dissection times.
  * Number of trocars.
  * Number of clips placed for the cystic duct and the cystic artery.
  * Rule of extraction of the gallbladder.
  * Use of antibiotics postoperatively.
  * Abdominal drainage.
  * length of hospital stay after surgery.
  To find a correlation between the variables of Group A and B, a test, a χ 2 tests were used to compare some surgical practices in different groups of surgeons, a (P < 0.05) was considered statistically significant.

IPD SHARING:
Plan to Share IPD: No